CLINICAL TRIAL: NCT01598753
Title: Phase 3 Double Blind Randomized Study Comparing Drug Treatment (Tramadol Versus Placebo) and Behavioral Health Treatments (Cognitive Behavioral Therapy Versus Health Education) for Patients With Fibromyalgia
Brief Title: Combined Behavioral and Analgesic Trial for Fibromyalgia
Acronym: COMBAT-FM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dennis Turk, Professor, Anesthesiology, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00001259
Record Dates: First submitted 2012-05-01; First posted 2012-05-15 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Tramadol; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tramadol (Active Comparator)
  Interventions: Drug: Tramadol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cognitive Behavior Therapy for FM (Active Comparator)
  Interventions: Behavioral: Cognitive Behavior Therapy for FM
- Health Education (Sham Comparator)
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Drug: Tramadol — 50 mg tablets titrated up to 2 tablets four times per day for a maximum dose of 400mg per day.
  Minimum accepted dose of 200mg per day
  Arms: Tramadol
Drug: Placebo — Pharmacological inactive tablet, 50mg tablets titrated to 2 tabs per day up to 400mg
  Arms: Placebo
Behavioral: Cognitive Behavior Therapy for FM — Subjects will be seen for 8 weekly 50 minute sessions of Cognitive Behavior Therapy that has been specifically tailored for Fibromyalgia patients.
  Arms: Cognitive Behavior Therapy for FM
Behavioral: Health Education — Subjects will receive 8 weekly 50 minute sessions of Health Education on Fibromyalgia
  Arms: Health Education

SUMMARY:
This is a randomized control study that involves a combination of a drug treatment, behavioral health, and placebo controls.

Some participants will receive a medication approved by the Food and Drug Administration for treatment of moderate to moderately severe pain called Tramadol HC1 IR. Others will receive an inactive pill, called a placebo. There will also be 2 different types of behavioral health treatments, Cognitive-Behavior Therapy (CBT) and Health Education (HE) both of which have been recommended for the treatment of patients with FM by the American Pain Society.

There are 4 possible study treatment combinations:

1. Tramadol + CBT,
2. Tramadol + HE,
3. Placebo + CBT,
4. Placebo + HE.

Although Tramadol, CBT, and HE have been shown to have some benefits for FM patients, there have been no studies that have evaluated the combination of medication and a behavioral health treatment. The primary purpose of this study is to compare the benefits of the 4 combinations listed.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 21-70
* Diagnosis of Fibromyalgia
* Current primary care physician
* Fluent in English

Exclusion Criteria:

* Rheumatologic disorders
* Drug and alcohol abuse in the past year
* Psychiatric hospitalization in the past 6 months
* Current use of Tramadol
* Certain antidepressant and other pain medications

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-05; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Rochester, Rochester, New York
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with fibromyalgia (FM) were enrolled at 2 sites, the University of Washington in Seattle WA and the University of Rochester in Rochester NY.
Pre-assignment Details: Participants underwent a physical exam to rule out conflicting medical conditions and confirm a diagnosis of FM (1990 ACR criteria). A 5-day baseline diary was distributed and required a mean daily pain score ≥ 4 and ≤ 9. A urine drug test with no illicit drugs and a negative urine pregnancy test (when applicable) were also required at baseline.
Groups:
- Placebo and Health Education: Participants received a matching placebo and 8 weekly 50 minute sessions of health education on Fibromyalgia.
- Tramadol and Health Education: Participants received between 200mg and 400mg of Tramadol daily and 8 weekly 50 minute sessions of health education on Fibromyalgia.
- Placebo and Cognitive Behavioral Therapy: Participants received matching placebo and 8 weekly 50 minute sessions of Cognitive Behavioral Therapy that had been specifically tailored for Fibromyalgia patients.
- Tramadol and Cognitive Behavioral Therapy: Participants received between 200mg and 400mg of Tramadol daily and 8 weekly 50 minute sessions of Cognitive Behavioral Therapy that had been specifically tailored for Fibromyalgia patients.
Period: Overall Study
Arm/Group | Placebo and Health Education | Tramadol and Health Education | Placebo and Cognitive Behavioral Therapy | Tramadol and Cognitive Behavioral Therapy
Started | 37 | 31 | 32 | 34
Completed | 25 | 16 | 24 | 19
Not Completed | 12 | 15 | 8 | 15
Not completed — Adverse Event | 1 | 9 | 1 | 7
Not completed — Lost to Follow-up | 4 | 3 | 7 | 5
Not completed — Physician Decision | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Health Education | Tramadol and Health Education | Placebo and Cognitive Behavioral Therapy | Tramadol and Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 37 | 31 | 32 | 34 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.9) | 51.2 (10.8) | 48.9 (13.1) | 44.64 (13.1) | 48.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 30 | 31 | 123
  Male | 3 | 3 | 2 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 1 | 6
  Not Hispanic or Latino | 36 | 29 | 30 | 33 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 35 | 25 | 29 | 28 | 117
  More than one race | 1 | 1 | 1 | 3 | 6
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 30% Improvement in Pain or 20% Improvement in Function
Description: The primary outcome is a reduction of at least 30% on the pain score (mean for 5-day daily pain diary) or improvement of 20% physical function (FIQR) from baseline (pre-treatment) to post-treatment. Individuals who achieve such decrease in pain or increase in function are labeled "responders."
Time Frame: Baseline (one week prior to drug titration) to post-treatment (approximately 11 weeks after baseline).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo and Health Education | Tramadol and Health Education | Placebo and Cognitive Behavioral Therapy | Tramadol and Cognitive Behavioral Therapy
Number analyzed (Participants) | 37 | 31 | 32 | 34
Participants | 24 | 13 | 21 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were reported from signing the informed consent until the completion of the 6-month follow-up visit.
Arm/Group | Placebo and Health Education | Tramadol and Health Education | Placebo and Cognitive Behavioral Therapy | Tramadol and Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/31 | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/31 | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 23/37 | 27/31 | 21/32 | 25/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Health Education (N=37) | Tramadol and Health Education (N=31) | Placebo and Cognitive Behavioral Therapy (N=32) | Tramadol and Cognitive Behavioral Therapy (N=34)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Skin abrasions (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood in stool (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurry vision (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bruise (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Change in respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (Endocrine disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 8 (8) | 0 (0) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 2 (2) | 1 (1)
Cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Decreased taste sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 4 (4) | 3 (3) | 4 (4)
Difficulty concentrating (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Difficulty swallowing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dissociative state (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0) | 4 (4)
Drowsiness (Nervous system disorders) | 0 (0) | 4 (4) | 3 (3) | 4 (4)
Dry eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dry nose (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extra emotional (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flu (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fogginess (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goosebumps (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 11 (12) | 2 (2) | 6 (6)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Endocrine disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Hypersensitivity to smell (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Increased irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thumb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left elbow mass resected (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Light headed (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 13 (16) | 4 (5) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pins and needles (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Poor balance (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Runny nose (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scalp lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sensitivity to noise (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shakiness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning pain through urethra (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shocking sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sweats (Endocrine disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Swelling (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thoughts of self mutilation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
TMJ pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremors (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Twitching (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vivid dreams (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1) | 4 (4)
Wisdom tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Yeast infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT01598753/Prot_SAP_002.pdf